CLINICAL TRIAL: NCT04756700
Title: Validation of DigiCog (BCCAMS App) and Konectom™ Tools, for Supporting Digitalized Clinical Assessment of Cognitive and Motor Functions in Patients With Multiple Sclerosis. DigiToms Study
Brief Title: Validation of DigiCog and Konectom Tools to Support Digitalized Clinical Assessment in Multiple Sclerosis
Acronym: DigiToms
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Biogen (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: FR-MSG-11654; 2020-A01801-38 (Other: ANSM)
Record Dates: First submitted 2021-02-12; First posted 2021-02-16 (Actual); Last update posted 2023-04-18 (Actual); Status verified 2023-04

CONDITIONS: Multiple Sclerosis
MeSH Terms: conditions — Multiple Sclerosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Healthy Participants (Experimental): Healthy participants matched with PwMS will have their cognitive and motor functions assessed using the DigiCog (BCCAMS app) tablet once in clinic and Konectom smartphone-based application for 2 days in clinic and at least 15 days at home.
  Interventions: Diagnostic Test: DigiCog (BCCAMS app); Diagnostic Test: Konectom Application
- PwMS: Participants with MS (Experimental): Participants with MS will have their cognitive and motor functions assessed using the DigiCog (BCCAMS app) tablet once in clinic and Konectom smartphone-based application for 2 days in clinic and at least 15 days at home.
  Interventions: Diagnostic Test: DigiCog (BCCAMS app); Diagnostic Test: Konectom Application

INTERVENTIONS:
Diagnostic Test: DigiCog (BCCAMS app) — Administered as specified in the treatment arm.
Diagnostic Test: Konectom Application — Administered as specified in the treatment arm.

SUMMARY:
The primary objective of this study is to establish scores of Cognitive impairment (CI) of the 3 DigiCog [Brief Computerized Cognitive Assessment for Multiple Sclerosis (BCCAMS) app] tests [Computerized Speed Cognitive Test (CSCT), Computerized Episodic Visual Memory Test (CEVMT) and the French Learning Test (FLT), a verbal memory test similar to the CVLT], using a tablet application in a sample of healthy participants matched to persons with MS (PwMS).

The secondary objectives of this study are to determine the ability of the DigiCog app to detect cognitive impairment (CI) compared to the classical Brief International Cognitive Assessment for MS (BICAMS) in PwMS; to determine the relationship between depressive symptoms and cognitive performance in Multiple Sclerosis (MS) sample; to determine the relationship between subjective perception of CI and cognitive performance ; to evaluate the reliability of Konectom™ digital outcome assessments (DOAs) in healthy subjects (HS) and PwMS; to evaluate the convergent validity of Konectom™ digital outcome assessments (DOAs) against in-clinic conventional disability outcome assessments in PwMS; to evaluate differences in Konectom™ DOAs [self administered at home and in-clinic] between PwMS and HS; to evaluate the variability of Konectom™ DOAs self-administered at home in free-living environment in HS and PwMS; to compare Konectom™ DOAs between in-clinic supervised administration versus self-assessments in free-living environment in HS and PwMS; to evaluate the clinical meaningfulness of Konectom™ DOAs against Patient-Reported Outcomes (PRO) in PwMS.

ELIGIBILITY:
Inclusion Criteria:

For PwMS:

* Expanded Disability Status Scale (EDSS) score ≤ 6.
* Multiple Sclerosis (MS) diagnosis according to 2017 revised McDonald criteria.

For Healthy Participants:

- Gender-, age- and education-matched with Multiple Sclerosis participants.

Exclusion Criteria:

For PwMS:

* Severe depression according to Diagnostic and Statistical Manual of Mental Disorders-5 (DSM-5) classification or severe on-going psychiatric condition, as per evaluation by the investigator;
* Change of Disease Modifiying Treatment (DMT) in the last 1 month;
* Any clinically significant neurological disorders other than MS, as per evaluation by the investigator;
* Any change of psychotropic treatment in the last 1 month;
* Clinically significant addiction (alcohol or other drug abuse), as per evaluation by the investigator;
* Recent acute relapse or disability worsening (less than one month);
* Steroid course in the previous month;
* Neuropsychological testing with the following tests in the previous year: Full BICAMS or DigiCog (BCCAMS app) battery, Fatigue Scale for Motor and Congnitive functions (FSMC), Computerized speed cognitive test (CSCT), Computerized Episodic Visual Memory Test (CEVMT), French Learning Test (FLT), Cognitive processing speed (CPS), Symbol Digit Modalities Test (SDMT);
* Developmental learning disabilities, as per evaluation by the investigator;
* Pregnant or breastfeeding women

For Health Participants:

* Severe depression (according to DSM-5 classification) or severe on-going psychiatric condition, as per evaluation by the investigator;
* Any clinically significant neurological disorders, as per evaluation by the investigator;
* Any psychotropic therapy consumption;
* Clinically significant addiction (alcohol or other drug abuse), as per evaluation by the investigator;
* Clinically significant cognitive complaint(s), as per evaluation by the investigator;
* Previous participation in other cognitive study using the same tests (Full BICAMS or DigiCog (BCCAMS app) battery, Fatigue Scale for Motor and Congnitive functions (FSMC), Computerized speed cognitive test (CSCT), Computerized Episodic Visual Memory Test (CEVMT), French Learning Test (FLT), Cognitive processing speed (CPS), Symbol Digit Modalities Test (SDMT));
* Developmental learning disabilities, as per evaluation by the investigator;
* Pregnant or breastfeeding women.

NOTE: Other protocol defined inclusion/ exclusion criteria may apply.

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 158 (Actual)
Dates: Start 2020-10-12 (Actual); Primary Completion 2022-07-26 (Actual); Study Completion 2022-07-26 (Actual)

PRIMARY OUTCOMES:
Raw Score of the Computerized Speed Cognitive Test (CSCT) using DigiCog (BCCAMS app) | Up to Day 28
  Number of the correct answers will provide raw score of CSCT from which regression based norms will be calculated.
Raw Score of the Computerized Episodic Visual Memory Test (CEVMT) using DigiCog (BCCAMS app) | Up to Day 28
  Total number of correct answers of the 3 trials will provide raw score of CEVMT from which regression based norms will be calculated.
Raw Score of the French Learning Test (FLT), using DigiCog (BCCAMS app) | Up to Day 28
  Total number of correct answers for the 5 trials will provide raw score of FLT from which regression based norms will be calculated.

SECONDARY OUTCOMES:
Sensitivity of the DigiCog (BCCAMS app) to detect CI in PwMS as compared to the Brief International Cognitive Assessment for MS (BICAMS) | Up to Day 28
  CI will be defined for DigiCog (BCCAMS app) as one or more abnormal test within the MS sample for DigiCog (BCCAMS app) as well as the BICAMS.
  The reference will be CI defined as one or more abnormal BICAMS test.
Specificity of the DigiCog (BCCAMS app) to detect CI in PwMS as compared to the BICAMS | Up to Day 28
  CI will be defined for DigiCog (BCCAMS app) as one or more abnormal test within the MS sample for DigiCog (BCCAMS app) as well as the BICAMS.
  The reference will be CI defined as one or more abnormal BICAMS test.
Accuracy of the DigiCog (BCCAMS app) to detect CI in PwMS as compared to the BICAMS | Up to Day 28
  CI will be defined for DigiCog (BCCAMS app) as one or more abnormal test within the MS sample for DigiCog (BCCAMS app) as well as the BICAMS.
  The reference will be CI defined as one or more abnormal BICAMS test.
Relationship between Depressive Symptoms with BDI FAST and Cognitive Performance ((BICAMS/DigiCog) | Up to Day 28
  Depressive symptoms will be estimated by BDI FAST (depressive scale) score. The BICAMS is used as the reference for the cognitive performances. The BCCAMS app is evaluated by using DigiCog scores.
Relationship Between Subjective Perception of CI with DailyCog and Cognitive Performance (BICAMS/DigiCog) | Up to Day 28
  Subjective perception of CI will be estimated by Daily Cog score. The BICAMS is used as the reference for the cognitive performances.
Reliability of Konectom Digital Outcome Assessment (DOA) in HS and PwMS: Intraclass Correlation Coefficient (ICC) of the score for Cognitive Processing Speed test (CPS) | Up to Day 28
Reliability of Konectom DOA in HS and PwMS: ICC of the score for Pinching Test | Up to Day 28
Reliability of Konectom DOA HS and PwMS: ICC of the score for Drawing Test | Up to Day 28
Reliability of Konectom DOA HS and PwMS: ICC of the score for Grip Force Tests | Up to Day 28
Reliability of Konectom DOA in HS and PwMS: ICC of the score for 6-minute Walk Test (6MWT) | Up to Day 28
Reliability of Konectom DOA in HS and PwMS: ICC of the score for U-turn Test (UTT) | Up to Day 28
Reliability of Konectom DOA in HS and PwMS: ICC of the score for Static Balance test (SBT) | Up to Day 28
Convergent Validity of Konectom DOA Against In-clinic Conventional Disability Outcome Assessment: CPS Versus Symbol Digit Modalities Test (SDMT) in PwMS | Up to Day 28
Convergent Validity of Konectom DOA Against In-clinic Conventional Disability Outcome Assessment: Pinching Versus 9-Hole Peg Test (9HPT) in PwMS | Up to Day 28
Convergent Validity of Konectom DOA Against In-clinic Conventional Disability Outcome Assessment: Drawing Versus 9HPT in PwMS | Up to Day 28
Convergent Validity of Konectom DOA Against In-clinic Conventional Disability Outcome Assessment: Grip Force Test Versus 9HPT in PwMS | Up to Day 28
Convergent Validity of Konectom DOA Against In-clinic Conventional Disability Outcome Assessment: SBT Versus Timed 25-foot Walk Test (T25FW) in PwMS | Up to Day 28
Convergent Validity of Konectom DOA Against In-clinic Conventional Disability Outcome Assessment: UTT Versus T25FW in PwMS | Up to Day 28
Convergent Validity of Konectom DOA Against In-clinic Conventional Disability Outcome Assessment: 6MWT Versus T25FW in PwMS | Up to Day 28
Convergent Validity of Konectom DOA Against In-clinic Conventional Disability Outcome Assessment: Passive Mobility Versus T25FW in PwMS | Up to Day 28
Convergent Validity of Konectom DOA Against In-clinic Conventional Disability Outcome Assessment: Konectom™ overall disability Versus Expanded Disability Status Scale (EDSS) and its Subscores in PwMS | Up to Day 28
Difference in Konectom DOA (Self-administered at Home and In-clinic) Between PwMS and HS: CPS Score | Up to Day 28
  Difference between PwMS and HS in the scores of CPS test during each testing condition will be evaluated.
Difference in Konectom DOA (Self-administered at Home and In-clinic) Between PwMS and HS: Pinching Test Score | Up to Day 28
  Difference between PwMS and HS in the score of pinching test during each testing condition will be evaluated
Difference in Konectom DOA (Self-administered at Home and In-clinic) Between PwMS and HS: Drawing Test Score | Up to Day 28
  Difference between PwMS and HS in the score of drawing test during each testing condition will be evaluated.
Difference in Konectom DOA (Self-administered at Home and In-clinic) Between PwMS and HS: Grip Force Test Score | Up to Day 28
  Difference between PwMS and HS in the score of grip force test during each testing condition will be evaluated.
Difference in Konectom DOA (Self-administered at Home and In-clinic) Between PwMS and HS: 6MWT Score | Up to Day 28
  Difference between PwMS and HS in the score of 6MWT test during each testing condition will be evaluated.
DDifference in Konectom DOA (Self-administered at Home and In-clinic) Between PwMS and HS: UTT Score | Up to Day 28
  Difference between PwMS and HS in the score of UTT test during each testing condition will be evaluated.
Difference in Konectom DOA (Self-administered at Home and In-clinic) Between PwMS and HS: SBT Score | Up to Day 28
  Difference between PwMS and HS in the score of SBT test during each testing condition will be evaluated.
Difference in Konectom DOA (Self-administered at Home and In-clinic) Between PwMS and HS: Mobility Behavior Score | Up to Day 28
  Difference between PwMS and HS in the score of mobility behavior test during each testing condition will be evaluated.
Difference in Konectom DOA (Self-administered at Home and In-clinic) Between PwMS and HS: Mood Scale Question (MSQ) | Up to Day 28
Variability of the Participant Performance throughout Konectom™ DOAs Self-administered at Home in Free-living Environment in HS and PwMS: CPS Score | Up to Day 28
Variability of the Participant Performance throughout Konectom™ DOAs Self-administered at Home in Free-living Environment in HS and PwMS: Pinching Test Score | Up to Day 28
Variability of the Participant Performance throughout Konectom™ DOAs Self-administered at Home in Free-living Environment in HS and PwMS: Drawing Test Score | Up to Day 28
Variability of the Participant Performance throughout Konectom™ DOAs Self-administered at Home in Free-living Environment in HS and PwMS: Grip Force Test Score | Up to Day 28
Variability of the Participant Performance throughout Konectom™ DOAs Self-administered at Home in Free-living Environment in HS and PwMS: 6MWT Score | Up to Day 28
Variability of the Participant Performance throughout Konectom™ DOAs Self-administered at Home in Free-living Environment in HS and PwMS: UTT Score | Up to Day 28
Variability of the Participant Performance throughout Konectom™ DOAs Self-administered at Home in Free-living Environment in HS and PwMS: SBT Score | Up to Day 28
Difference in Konectom DOA Between In-clinic Supervised Administration Versus Self-assessments in Free-living Environment in HS and PwMS | Up to Day 28
Clinical Meaningfulness of Konectom DOA Against PRO: CPS Association with Cognitive Sub-Scores of the Fatigue Scale for Motor and Cognitive Functions (FSMC) in PwMS | Up to Day 28
Clinical Meaningfulness of Konectom DOA Against PRO: CPS Association with Cognitive/Psychological Items of the Multiple Sclerosis Impact Scale 29 (MSIS-29) in PwMS | Up to Day 28
Clinical Meaningfulness of Konectom DOA Against PRO: CPS Association with Daily Cog in PwMS | Up to Day 28
Clinical Meaningfulness of Konectom DOA Against PRO: Pinching Test Association with ABILHAND-56 in PwMS | Up to Day 28
Clinical Meaningfulness of Konectom DOA Against PRO: Pinching Test Association with early MS manual ability questionnaires | Up to Day 28
Clinical Meaningfulness of Konectom DOA Against PRO: Drawing Test Association with ABILHAND-56 in PwMS | Up to Day 28
Clinical Meaningfulness of Konectom DOA Against PRO: Drawing Test Association with early MS manual ability questionnaires | Up to Day 28
Clinical Meaningfulness of Konectom DOA Against PRO: Grip Force Test Association with ABILHAND-56 in PwMS | Up to Day 28
Clinical Meaningfulness of Konectom DOA Against PRO: Grip Force Test Association with Early MS Manual Ability Questionnaires | Up to Day 28
Clinical Meaningfulness of Konectom DOA Against PRO: SBT Association with Multiple Sclerosis Walking Scale 12 items (MSWS-12) in PwMS | Up to Day 28
Clinical Meaningfulness of Konectom DOA Against PRO: SBT Association with Early MS Walking Ability-gait Questionnaires in PwMS | Up to Day 28
Clinical Meaningfulness of Konectom DOA Against PRO: SBT Association with Ambulation-related Items of the MSIS-29 in PwMS | Up to Day 28
Clinical Meaningfulness of Konectom DOA Against PRO: SBT Association with PDDS in PwMS | Up to Day 28
Clinical Meaningfulness of Konectom DOA Against PRO: UTT Association with MSWS-12 in PwMS | Up to Day 28
Clinical Meaningfulness of Konectom DOA Against PRO: UTT Association with Early MS Walking Ability-gait Questionnaires in PwMS | Up to Day 28
Clinical Meaningfulness of Konectom DOA Against PRO: UTT Association with Ambulation-related Items of the MSIS-29 in PwMS | Up to Day 28
Clinical Meaningfulness of Konectom DOA Against PRO: UTT Association with PDDS in PwMS | Up to Day 28
Clinical Meaningfulness of Konectom DOA Against PRO: 6MWT Association with MSWS-12 in PwMS | Up to Day 28
Clinical Meaningfulness of Konectom DOA Against PRO: 6MWT Association with Early MS Walking Ability-gait Questionnaires in PwMS | Up to Day 28
Clinical Meaningfulness of Konectom DOA Against PRO: 6MWT Association with Ambulation-related Items of the MSIS-29 in PwMS | Up to Day 28
Clinical Meaningfulness of Konectom DOA Against PRO: 6MWT Association with PDDS in PwMS | Up to Day 28
Clinical Meaningfulness of Konectom DOA Against PRO: Passive Mobility Association with MSWS-12 in PwMS | Up to Day 28
Clinical Meaningfulness of Konectom DOA Against PRO: Passive Mobility Association with Early MS Walking Ability-gait Questionnaires in PwMS | Up to Day 28
Clinical Meaningfulness of Konectom DOA Against PRO: Passive Mobility Association with Ambulation-related Items of the MSIS-29 in PwMS | Up to Day 28
Clinical Meaningfulness of Konectom DOA Against PRO: Passive Mobility Association with PDDS in PwMS | Up to Day 28

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Biogen
Locations (1):
- Research Site, Bordeaux, France

IPD SHARING:
Plan to Share IPD: Yes
In accordance with Biogen's Clinical Trial Transparency and Data Sharing Policy on https://www.biogentrialtransparency.com/
URL: https://vivli.org/